CLINICAL TRIAL: NCT03422198
Title: Short Course Adjuvant Vaginal Cuff Brachytherapy (VCB) in Early Endometrial Cancer Compared to Standard of Care (SAVE)
Brief Title: Short Course Vaginal Cuff Brachytherapy in Treating Participants With Stage I-II Endometrial Cancer
Acronym: SAVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Huntsman Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI103841; NCI-2018-00011 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Endometrial Endometrioid Adenocarcinoma; Endometrial Serous Adenocarcinoma; Stage I Uterine Corpus Cancer; Stage IA Uterine Corpus Cancer; Stage IB Uterine Corpus Cancer; Stage II Uterine Corpus Cancer; Uterine Corpus Carcinosarcoma; Uterine Corpus Sarcoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Short course vaginal cuff brachytherapy (Experimental): Participants undergo short course vaginal cuff brachytherapy for 2 fractions with 1 week apart.
  Interventions: Radiation: Short course vaginal cuff brachytherapy
- Vaginal cuff brachytherapy (Active Comparator): Participants undergo standard of care vaginal cuff brachytherapy for 3-5 fractions over no more than 3 weeks.
  Interventions: Radiation: Vaginal Cuff Brachytherapy

INTERVENTIONS:
Radiation: Vaginal Cuff Brachytherapy — Undergo standard of care vaginal cuff brachytherapy
  Other Names: best practice; standard of care; standard therapy
  Arms: Vaginal cuff brachytherapy
Radiation: Short course vaginal cuff brachytherapy — Undergo short course vaginal cuff brachytherapy
  Other Names: BRACHYTHERAPY; internal radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy
  Arms: Short course vaginal cuff brachytherapy

SUMMARY:
This randomized phase III trial studies short course vaginal cuff brachytherapy to see how well it works compared with standard of care vaginal cuff brachytherapy in treating participants with stage I-II endometrial cancer. Short course vaginal cuff brachytherapy, also known as internal radiation therapy, uses (over a shorter period) radioactive material placed directly into or near a tumor in the upper portion of the vagina to kill tumor cells.

After completion of cohort 1 (108 participants), the protocol was expended to add a second cohort of 80 additional participants, and re-opened study recruitment.

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic cancer in the Western world and primarily affects postmenopausal women. The primary form of treatment is surgery, consisting of a total abdominal or laparoscopic hysterectomy and bilateral salpingo-oophorectomy. Adjuvant radiotherapy for endometrial cancer has been studied in prospective trials for at least four decades. All trials have demonstrated an improvement in local regional control. However, improvement in survival has not been observed in prospective randomized trials in early-stage patients.

There is great heterogeneity in prognoses in stage I patients. National Comprehensive Cancer Network (NCCN) guidelines consequently recommend no treatment in general for low-stage patients, adjuvant brachytherapy for patients with intermediate- and high-intermediate-risk disease, and for patients with deeply invasive tumors with high-grade lesions, external beam radiotherapy is an option (NCCN Guidelines 2016). Over the ensuing decades, there has been a shift toward increasing use of vaginal cuff brachytherapy.

This is a phase III, unblinded, randomized trial comparing an experimental arm and a control arm of vaginal cuff brachytherapy: The experimental arm will treat subjects with 2 fractions of vaginal brachytherapy. The control arm will treat subjects with standard-of-care vaginal cuff brachytherapy of 3-5 fractions. Patients will be randomized 1:1 to the different treatment arms.

After completion of cohort 1 (108 participants), the protocol was expanded to add a second cohort of 80 additional participants, and reopened study recruitment.

Cohort 1 evaluated the non-inferiority of patient Health Related Quality of Life (HRQOL) in the experimental arm compared to the control arm using the Global Health Status from the EORTC QLQ-C30. Cohort 2 will evaluate the frequency and severity of patient-reported financial toxicity in patients with early-stage endometrial cancer treated with vaginal cuff-brachytherapy (VCB) at one month post-VCB.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial carcinoma: endometrioid type, serous, and clear cell, to include tumors originating in the cervix, but are primarily located in the uterus, and for whom vaginal cuff brachytherapy is indicated. Carcinosarcoma and other sarcomas are permitted; Federation of Gynecology and Obstetrics (FIGO) stage I and stage II, with one of the following combinations of stage and grade:

  * Stage IA, grade 1 with LVSI, 2, 3
  * Stage IB, grades 1-3
  * Stage II, grades 1-3
  * Stage IIIA, grades 1-3, not receiving EBRT as part of adjuvant therapy.
* Participants post-hysterectomy and free from residual disease.
* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG)-performance status 0-2.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Life expectancy of >2 years.

Exclusion Criteria:

* Stages of endometrial carcinoma other than described.
* Previous pelvic radiotherapy.
* Concurrent malignancy requiring non-protocol anti-cancer treatment other than surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina DeCesaris, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (5):
- United States (5):
  - Stanford Cancer Center, Palo Alto, California
  - Loyola University Medical Center, Maywood, Illinois
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Intermountain Medical Center / LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pecorelli S. Revised FIGO staging for carcinoma of the vulva, cervix, and endometrium. Int J Gynaecol Obstet. 2009 May;105(2):103-4. doi: 10.1016/j.ijgo.2009.02.012. No abstract available. PMID 19367689
- [Background] Briet JM, Hollema H, Reesink N, Aalders JG, Mourits MJ, ten Hoor KA, Pras E, Boezen HM, van der Zee AG, Nijman HW. Lymphvascular space involvement: an independent prognostic factor in endometrial cancer. Gynecol Oncol. 2005 Mar;96(3):799-804. doi: 10.1016/j.ygyno.2004.11.033. PMID 15721428
- [Background] Cohn DE, Horowitz NS, Mutch DG, Kim SM, Manolitsas T, Fowler JM. Should the presence of lymphvascular space involvement be used to assign patients to adjuvant therapy following hysterectomy for unstaged endometrial cancer? Gynecol Oncol. 2002 Dec;87(3):243-6. doi: 10.1006/gyno.2002.6825. PMID 12468320
- [Background] Thomas GM. A role for adjuvant radiation in clinically early carcinoma of the endometrium? Int J Gynecol Cancer. 2010 Oct;20(11 Suppl 2):S64-6. doi: 10.1111/IGC.0b013e3181f5c688. PMID 20975365
- [Background] Bosse T, Peters EE, Creutzberg CL, Jurgenliemk-Schulz IM, Jobsen JJ, Mens JW, Lutgens LC, van der Steen-Banasik EM, Smit VT, Nout RA. Substantial lymph-vascular space invasion (LVSI) is a significant risk factor for recurrence in endometrial cancer--A pooled analysis of PORTEC 1 and 2 trials. Eur J Cancer. 2015 Sep;51(13):1742-50. doi: 10.1016/j.ejca.2015.05.015. Epub 2015 Jun 3. PMID 26049688
- [Background] Lee CM, Szabo A, Shrieve DC, Macdonald OK, Gaffney DK. Frequency and effect of adjuvant radiation therapy among women with stage I endometrial adenocarcinoma. JAMA. 2006 Jan 25;295(4):389-97. doi: 10.1001/jama.295.4.389. PMID 16434629
- [Background] Kirchheiner K, Czajka-Pepl A, Ponocny-Seliger E, Scharbert G, Wetzel L, Nout RA, Sturdza A, Dimopoulos JC, Dorr W, Potter R. Posttraumatic stress disorder after high-dose-rate brachytherapy for cervical cancer with 2 fractions in 1 application under spinal/epidural anesthesia: incidence and risk factors. Int J Radiat Oncol Biol Phys. 2014 Jun 1;89(2):260-7. doi: 10.1016/j.ijrobp.2014.02.018. Epub 2014 Apr 7. PMID 24721589
- [Background] Aalders J, Abeler V, Kolstad P, Onsrud M. Postoperative external irradiation and prognostic parameters in stage I endometrial carcinoma: clinical and histopathologic study of 540 patients. Obstet Gynecol. 1980 Oct;56(4):419-27. PMID 6999399
- [Background] Creutzberg CL, van Putten WL, Koper PC, Lybeert ML, Jobsen JJ, Warlam-Rodenhuis CC, De Winter KA, Lutgens LC, van den Bergh AC, van de Steen-Banasik E, Beerman H, van Lent M. Surgery and postoperative radiotherapy versus surgery alone for patients with stage-1 endometrial carcinoma: multicentre randomised trial. PORTEC Study Group. Post Operative Radiation Therapy in Endometrial Carcinoma. Lancet. 2000 Apr 22;355(9213):1404-11. doi: 10.1016/s0140-6736(00)02139-5. PMID 10791524
- [Background] Keys HM, Roberts JA, Brunetto VL, Zaino RJ, Spirtos NM, Bloss JD, Pearlman A, Maiman MA, Bell JG; Gynecologic Oncology Group. A phase III trial of surgery with or without adjunctive external pelvic radiation therapy in intermediate risk endometrial adenocarcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2004 Mar;92(3):744-51. doi: 10.1016/j.ygyno.2003.11.048. PMID 14984936
- [Background] ASTEC/EN.5 Study Group; Blake P, Swart AM, Orton J, Kitchener H, Whelan T, Lukka H, Eisenhauer E, Bacon M, Tu D, Parmar MK, Amos C, Murray C, Qian W. Adjuvant external beam radiotherapy in the treatment of endometrial cancer (MRC ASTEC and NCIC CTG EN.5 randomised trials): pooled trial results, systematic review, and meta-analysis. Lancet. 2009 Jan 10;373(9658):137-46. doi: 10.1016/S0140-6736(08)61767-5. Epub 2008 Dec 16. PMID 19070891
- [Background] Nout RA, Smit VT, Putter H, Jurgenliemk-Schulz IM, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Mens JW, Slot A, Kroese MC, van Bunningen BN, Ansink AC, van Putten WL, Creutzberg CL; PORTEC Study Group. Vaginal brachytherapy versus pelvic external beam radiotherapy for patients with endometrial cancer of high-intermediate risk (PORTEC-2): an open-label, non-inferiority, randomised trial. Lancet. 2010 Mar 6;375(9717):816-23. doi: 10.1016/S0140-6736(09)62163-2. PMID 20206777
- [Background] Nout RA, Putter H, Jurgenliemk-Schulz IM, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Mens JW, Slot A, Stenfert Kroese MC, van Bunningen BN, Smit VT, Nijman HW, van den Tol PP, Creutzberg CL. Quality of life after pelvic radiotherapy or vaginal brachytherapy for endometrial cancer: first results of the randomized PORTEC-2 trial. J Clin Oncol. 2009 Jul 20;27(21):3547-56. doi: 10.1200/JCO.2008.20.2424. Epub 2009 Jun 22. PMID 19546404
- [Background] Sorbe B, Straumits A, Karlsson L. Intravaginal high-dose-rate brachytherapy for stage I endometrial cancer: a randomized study of two dose-per-fraction levels. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1385-9. doi: 10.1016/j.ijrobp.2004.12.079. PMID 16029797
- [Background] McMeekin DS, The University of Oklahoma OC, OK, United States, Filiaci VL, et al. 1A randomized phase III trial of pelvic radiation therapy (PXRT) versus vaginal cuff brachytherapy followed by paclitaxel/carboplatin chemotherapy (VCB/C) in patients with high risk (HR), early stage endometrial cancer (EC): A Gynecologic Oncology Group trial. Gynecol Oncol. 2014;134: 438.
- [Background] Harkenrider MM, Block AM, Alektiar KM, Gaffney DK, Jones E, Klopp A, Viswanathan AN, Small W Jr. American Brachytherapy Task Group Report: Adjuvant vaginal brachytherapy for early-stage endometrial cancer: A comprehensive review. Brachytherapy. 2017 Jan-Feb;16(1):95-108. doi: 10.1016/j.brachy.2016.04.005. Epub 2016 May 31. PMID 27260082
- [Background] Delaney G, Jacob S, Barton M. Estimation of an optimal radiotherapy utilization rate for gynecologic carcinoma: part II--carcinoma of the endometrium. Cancer. 2004 Aug 15;101(4):682-92. doi: 10.1002/cncr.20445. PMID 15305397
- [Background] Lee CM, Szabo A, Shrieve DC, Macdonald OK, Tward JD, Skidmore TB, Gaffney DK. Descriptive nomograms of adjuvant radiotherapy use and patterns of care analysis for stage I and II endometrial adenocarcinoma: A surveillance, epidemiology, and end results population study. Cancer. 2007 Nov 1;110(9):2092-100. doi: 10.1002/cncr.22997. PMID 17849468
- [Background] Punglia RS, Weeks JC, Neville BA, Earle CC. Effect of distance to radiation treatment facility on use of radiation therapy after mastectomy in elderly women. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):56-63. doi: 10.1016/j.ijrobp.2006.03.059. Epub 2006 Jul 11. PMID 16814955
- [Background] Scott NW, Fayers PM, Aaronson NK et al (2008) EORTC QLQ-C30 Reference Values. European Organization for Research and Treatment of Cancer.
- [Background] Cocks K, King MT, Velikova G, Fayers PM, Brown JM. Quality, interpretation and presentation of European Organisation for Research and Treatment of Cancer quality of life questionnaire core 30 data in randomised controlled trials. Eur J Cancer. 2008 Sep;44(13):1793-8. doi: 10.1016/j.ejca.2008.05.008. Epub 2008 Jul 1. PMID 18599286
- [Background] Maringwa JT, Quinten C, King M, Ringash J, Osoba D, Coens C, Martinelli F, Vercauteren J, Cleeland CS, Flechtner H, Gotay C, Greimel E, Taphoorn MJ, Reeve BB, Koch JS, Weis J, Smit EF, van Meerbeeck JP, Bottomley A; EORTC PROBE project and the Lung Cancer Group. Minimal important differences for interpreting health-related quality of life scores from the EORTC QLQ-C30 in lung cancer patients participating in randomized controlled trials. Support Care Cancer. 2011 Nov;19(11):1753-60. doi: 10.1007/s00520-010-1016-5. Epub 2010 Oct 1. PMID 20886240
- [Background] Zafar SY, Peppercorn JM, Schrag D, Taylor DH, Goetzinger AM, Zhong X, Abernethy AP. The financial toxicity of cancer treatment: a pilot study assessing out-of-pocket expenses and the insured cancer patient's experience. Oncologist. 2013;18(4):381-90. doi: 10.1634/theoncologist.2012-0279. Epub 2013 Feb 26. PMID 23442307
- [Background] Neugut AI, Subar M, Wilde ET, Stratton S, Brouse CH, Hillyer GC, Grann VR, Hershman DL. Association between prescription co-payment amount and compliance with adjuvant hormonal therapy in women with early-stage breast cancer. J Clin Oncol. 2011 Jun 20;29(18):2534-42. doi: 10.1200/JCO.2010.33.3179. Epub 2011 May 23. PMID 21606426
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Bouberhan S, Shea M, Kennedy A, Erlinger A, Stack-Dunnbier H, Buss MK, Moss L, Nolan K, Awtrey C, Dalrymple JL, Garrett L, Liu FW, Hacker MR, Esselen KM. Financial toxicity in gynecologic oncology. Gynecol Oncol. 2019 Jul;154(1):8-12. doi: 10.1016/j.ygyno.2019.04.003. Epub 2019 Apr 30. PMID 31053404
- [Background] Liang MI, Summerlin SS, Blanchard CT, Boitano TKL, Huh WK, Bhatia S, Pisu M. Measuring Financial Distress and Quality of Life Over Time in Patients With Gynecologic Cancer-Making the Case to Screen Early in the Treatment Course. JCO Oncol Pract. 2021 Oct;17(10):e1576-e1583. doi: 10.1200/OP.20.00907. Epub 2021 Feb 17. PMID 33596114
- [Background] Soisson S, Ganz PA, Gaffney D, Rowe K, Snyder J, Wan Y, Deshmukh V, Newman M, Fraser A, Smith K, Herget K, Hanson HA, Wu YP, Stanford J, Al-Sarray A, Werner TL, Setiawan VW, Hashibe M. Long-term Cardiovascular Outcomes Among Endometrial Cancer Survivors in a Large, Population-Based Cohort Study. J Natl Cancer Inst. 2018 Dec 1;110(12):1342-1351. doi: 10.1016/j.ygyno.2017.12.025. PMID 29741696
- [Background] Lee E, Zhu J, Velazquez J, Bernardo R, Garcia J, Rovito M, Hines RB. Evaluation of Diet Quality Among American Adult Cancer Survivors: Results From 2005-2016 National Health and Nutrition Examination Survey. J Acad Nutr Diet. 2021 Feb;121(2):217-232. doi: 10.1016/j.jand.2020.08.086. Epub 2020 Nov 3. PMID 33158797
- [Background] Smits A, Lopes A, Das N, Bekkers R, Massuger L, Galaal K. The effect of lifestyle interventions on the quality of life of gynaecological cancer survivors: A systematic review and meta-analysis. Gynecol Oncol. 2015 Dec;139(3):546-52. doi: 10.1016/j.ygyno.2015.10.002. Epub 2015 Oct 9. PMID 26441008
- [Background] Friedenreich CM, Cook LS, Wang Q, Kokts-Porietis RL, McNeil J, Ryder-Burbidge C, Courneya KS. Prospective Cohort Study of Pre- and Postdiagnosis Physical Activity and Endometrial Cancer Survival. J Clin Oncol. 2020 Dec 1;38(34):4107-4117. doi: 10.1200/JCO.20.01336. Epub 2020 Oct 7. PMID 33026939
- [Background] Kitson S, Ryan N, MacKintosh ML, Edmondson R, Duffy JM, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2018 Feb 1;2(2):CD012513. doi: 10.1002/14651858.CD012513.pub2. PMID 29388687
- [Background] Diet History Questionnaire III (DHQ III) | EGRP/DCCPS/NCI/NIH. Accessed October 29, 2022. https://epi.grants.cancer.gov/dhq3/
- [Background] Krebs-Smith SM, Pannucci TE, Subar AF, Kirkpatrick SI, Lerman JL, Tooze JA, Wilson MM, Reedy J. Update of the Healthy Eating Index: HEI-2015. J Acad Nutr Diet. 2018 Sep;118(9):1591-1602. doi: 10.1016/j.jand.2018.05.021. PMID 30146071

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Short Course Vaginal Cuff Brachytherapy: Participants undergo short course vaginal cuff brachytherapy for 2 fractions with 1 week apart.
- Control: Standard of Care Vaginal Cuff Brachytherapy: Participants undergo standard of care vaginal cuff brachytherapy for 3-5 fractions over no more than 3 weeks.
Period: Overall Study
Arm/Group | Experimental: Short Course Vaginal Cuff Brachytherapy | Control: Standard of Care Vaginal Cuff Brachytherapy
Started | 54 | 54
Completed | 54 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Short Course Vaginal Cuff Brachytherapy | Control: Standard of Care Vaginal Cuff Brachytherapy | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 31 | 53
  >=65 years | 32 | 23 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.31 (10.25) | 63.65 (9.68) | 64.48 (9.95)
Age, Continuous [Median (Full Range); unit: years] | 66.5 [40 to 84] | 63.5 [30 to 87] | 65 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 46 | 48 | 94
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 41 | 45 | 86
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 7 | 2 | 9
Baseline EORTC Quality of Life Score [Mean (Standard Deviation); unit: score on a scale] — The European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-30 (QLQ-30) is used to evaluate quality of life in cancer patients. The quality of life score ranges from 0-100, with higher scores indicating better quality of life. Population: The primary outcome related to this baseline measure requires participants to have completed both the baseline and Month 1 assessments to be included. Participants without both were excluded in this baseline measure. Five control arm participants did not complete the Month 1 questionnaire. One control arm participant did not complete the baseline questionnaire. Two experimental arm participants did not complete the Month 1 questionnaire.
  score on a scale
    number analyzed (Participants) | 52 | 48 | 100
    (all) | 72.28 (21.5) | 67.88 (21.74) | 70.17 (21.26)
Baseline EORTC Symptom Score [Mean (Standard Deviation); unit: score on a scale] — The European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Endometrial-24 (QLQ-EN24) was used to evaluate quality of life in cancer patients with endometrial cancers. From this assessment, one question was selected as an indicator for this outcome, which measured whether participants felt less feminine as a result of their disease or treatment. The score ranges from 0-100, with higher scores indicating feeling less feminine. Population: The secondary outcome related to this baseline measure requires participants to have completed both baseline and Month 1 questionnaires to be included. Participants who did not complete both were excluded. Five control arm participants did not complete the Month 1 questionnaire. One control arm participant did not complete the baseline questionnaire. Three experimental arm participants did not complete the Month 1 questionnaire.
  score on a scale
    number analyzed (Participants) | 51 | 48 | 99
    (all) | 10.46 (26.24) | 16.67 (28.35) | 13.47 (27.32)

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life From Baseline to 1 Month
Description: The European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-30 (QLQ-30) is used to evaluate quality of life in cancer patients. The questionnaire was given before and one month following treatment. The quality of life score ranges from 0-100, with higher scores indicating better quality of life. Baseline scores can be found in the Baseline Characteristics module. This outcome reports the average change from baseline to Month 1.
Time Frame: At 1 month post treatment
Population: Five control arm participants were excluded from analysis because they did not complete the Month 1 questionnaire. One control arm participant was excluded because they did not complete the baseline questionnaire. Two experimental arm participants were excluded from analysis because they did not complete the Month 1 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Short Course Vaginal Cuff Brachytherapy | Control: Standard of Care Vaginal Cuff Brachytherapy
Number analyzed (Participants) | 52 | 48
score on a scale | 2.08 (15.02) | 2.08 (18.23)

2. Primary Outcome: Cohort 2: Participant-Reported Financial Toxicity
Description: One month post-brachytherapy, participants will be given the Functional Assessment of Chronic Illness Therapy (FACIT) - COmprehensive Score for financial Toxicity (COST) (FACIT-COST) questionnaire. The score range is 0-44, with higher scores indicating better financial well-being. Mean scores will be reported.
Time Frame: One month after brachytherapy
Reporting Status: Not Posted

3. Secondary Outcome: Treatment-related Symptoms on HRQOL Using European Organization for Research and Treatment of Cancer Endometrial Cancer Module (EORTC EN24), Question 48
Description: The European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Endometrial-24 (QLQ-EN24) was used to evaluate quality of life in cancer patients with endometrial cancers. The questionnaire was given before and one month following treatment. From this assessment, one question was selected as an indicator for this outcome, which measured whether participants felt less feminine as a result of their disease or treatment. The score ranges from 0-100, with higher scores indicating feeling less feminine. Baseline scores can be found in the Baseline Characteristics module. This outcome reports the average change from baseline to Month 1.
Time Frame: one month post-treatment
Population: Five control arm participants were excluded from analysis because they did not complete the Month 1 questionnaire. One control arm participants was excluded because they did not complete the baseline questionnaire. Three experimental arm participants were excluded from analysis because they did not complete the Month 1 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Short Course Vaginal Cuff Brachytherapy | Control: Standard of Care Vaginal Cuff Brachytherapy
Number analyzed (Participants) | 51 | 48
score on a scale | 0.65 (22.6) | -6.25 (29.7)

4. Secondary Outcome: USD Amount Charged for Procedures
Description: The amount charged to participants or their insurance in US Dollars (USD) was collected to evaluate cost of experimental versus standard of care courses of treatment. Data was collected at approximately six months after treatment.
Time Frame: Approximately 6 months after treatment
Population: Amount charged for procedures could not be obtained for six participants on the experimental arm.
Measure: Mean (Standard Deviation); unit: US Dollars (USD)
Arm/Group | Experimental: Short Course Vaginal Cuff Brachytherapy | Control: Standard of Care Vaginal Cuff Brachytherapy
Number analyzed (Participants) | 48 | 54
US Dollars (USD) | 33204.97 (16867.76) | 45919.55 (19808.48)

5. Secondary Outcome: Cohort 2: Participant-Reported Diet
Description: Participants will be asked to complete the National Cancer Institute (NCI) Diet History Questionnaire 3 (DHQIII) through the NCI website. Additional information about the questionnaire, methods, and measurements will be updated when results are reported for this outcome.
Time Frame: One month after brachytherapy
Reporting Status: Not Posted

6. Secondary Outcome: Cohort 2: Participant-Reported Activity Levels
Description: Participants will be asked to complete the NCI Activities Completed over Time in 24-hours (ACT24) questionnaire through the NCI website. Additional information about the questionnaire, methods, and measurements will be updated when results are reported for this outcome.
Time Frame: One month after brachytherapy
Reporting Status: Not Posted

7. Secondary Outcome: Cohort 2: Financial Toxicity Correlated With Quality of Life
Description: Mean scores from the FACIT-COST (from Outcome Measure 2: Participant-Reported Financial Toxicity) will be correlated with mean QoL scores (from Outcome Measure 1). Additional information about the methods and measurements will be updated when results are reported for this outcome.
Time Frame: One month after brachytherapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months after start of brachytherapy
Description: Routine safety and tolerability were evaluated at each study visit from the results of reported signs and symptoms, scheduled physical examinations, vital sign measurements, and clinical laboratory test results. Information about all adverse events, whether volunteered by the participant, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, was collected, recorded and followed as appropriate.
Arm/Group | Experimental: Short Course Vaginal Cuff Brachytherapy | Control: Standard of Care Vaginal Cuff Brachytherapy
All-Cause Mortality (participants affected / at risk) | 2/54 | 1/54
Serious Adverse Events (participants affected / at risk) | 2/54 | 2/54
Other Adverse Events (participants affected / at risk) | 46/54 | 50/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Short Course Vaginal Cuff Brachytherapy (N=54) | Control: Standard of Care Vaginal Cuff Brachytherapy (N=54)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Short Course Vaginal Cuff Brachytherapy (N=54) | Control: Standard of Care Vaginal Cuff Brachytherapy (N=54)
Abdominal Distension (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 9 (10)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (4) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (6) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (14) | 16 (22)
Dizziness (Nervous system disorders) | 2 (2) | 3 (4)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 5 (5) | 4 (4)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fatigue (General disorders) | 20 (23) | 23 (29)
Fecal incontinence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (4) | 5 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1)
Generalized edema (General disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (2) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 2 (2)
INR increased (Investigations) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (4)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 9 (11)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (5) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 8 (9)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 9 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4 (4) | 4 (4)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 3 (3) | 5 (6)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 4 (4) | 10 (11)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (9)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (2) | 4 (4)
Vaginal discharge (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 4 (4) | 4 (5)
Vaginal hemorrhage (Reproductive system and breast disorders) | 4 (5) | 8 (8)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal pain (Reproductive system and breast disorders) | 4 (4) | 5 (5)
Vaginal stricture (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vulval infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 2 (2)
Weight loss (Investigations) | 1 (1) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03422198/Prot_SAP_001.pdf